CLINICAL TRIAL: NCT03147235
Title: The Effects of a Music Therapist Designed Listening Program on Intraoperative Vitrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Stephen J. Kim, MD, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #170400
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative; Music Therapy
MeSH Terms: conditions — Pain, Postoperative | interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitrectomy with music listening (Experimental): Patients undergoing vitrectomy surgery will listen to a designed playlist of music during the entire duration of surgery
  Interventions: Behavioral: vitrectomy with music listening
- vitrectomy without music listening (No Intervention): Patients undergoing vitrectomy surgery will not be exposed to music listening.

INTERVENTIONS:
Behavioral: vitrectomy with music listening — Those randomized to music listening will be exposed to a standardized playlist of previously validated relaxation music.
  Arms: vitrectomy with music listening

SUMMARY:
This will be a prospective, randomized controlled trial with patients randomly assigned to either the experimental or control group. The experimental group will be exposed to the independent variable (IV) and the control group will not be exposed to the IV. The IV will be a music therapist- designed listening program during surgery. A total of 60 patients will be consecutively enrolled and undergo block randomization to either a music listening group or a control group (no music). Trained medical research personnel will assist with various parts of the study and will be defined as those individuals who have completed and are up-to-date on the Collaborative Institutional Training Initiative (CITI) training. These individuals will consist of a board certified music therapist, practicing ophthalmologists, and physicians-in-training.

DETAILED DESCRIPTION:
This prospective trial will block randomize a consecutive cohort of patients undergoing routine vitrectomy surgery at an university hospital to a designed listening program during surgery or to nothing in order to determine whether music listening during surgery can measurably result in decreased patient pain assessed by the Wong-Baker Faces Pain scale. Secondary outcome measures will be blood pressure, need for anxiety medication, postoperative pain medication, and patient overall experience.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will consist of patients already scheduled for elective vitrectomy surgery at a tertiary academic university hospital.

Exclusion Criteria:

* Exclusion criteria consist of: patients with deafness or unilateral or bilateral severe hearing loss, unwillingness or inability to complete post-surgical surveys, previous vitrectomy surgeries, diagnosed anxiety disorder (claustrophobia, etc.), and/or chronic narcotic or substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
post-operative pain | during post-operative recovery time, approximately 2 hours
  post-operative pain as measured by the Wong-Baker Faces pain scale, 0 is no pain, 10 is the worst pain

SECONDARY OUTCOMES:
patient satisfaction | during postoperative recovery time, approximately 2 hours
  patient satisfaction as measured by a modified version of the The Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey
anti-anxiety medication | start to finish of surgery, approximately 1.5 hours
  amount of anti-anxiety medication administered during surgery
pain médication | start to finish of surgery, approximately 1.5 hours
  amount of pain medication administered during surgery
blood pressure | start to finish of surgery, approximately 1.5 hours
  blood pressure during the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kim, MD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No